CLINICAL TRIAL: NCT00005551
Title: Sleep Apnea in a Non-Clinical Population
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5095; R03HL062686 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes; Obesity; Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes; Obesity; Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To investigate the causes, consequences and quantitation of sleep disordered breathing (SDB).

DETAILED DESCRIPTION:
BACKGROUND:

The study utilized an extremely rich source of data collected on the Wisconsin Sleep Cohort, one of the largest cohort studies of SDB and one with the longest periods of follow-up, to address a broad array of questions related to the pathogenesis and risk of SDB in the general community. The data-set was obtained between 1988 and 1998 in a population of 1400 workers age 30 to 60 years, including an overnight sleep polysomnographic in-lab study conducted on two occasions over an eight year period. The dataset contained a computerized analysis of over 300,000 apneas and hypopneas in this non-clinical population.

Although strong associations have been demonstrated between sleep disordered breathing and cardiovascular diseases, much is not known regarding the mechanisms by which SDB produces blood pressure changes and increases morbidity. Further analysis of the polysomnography and blood pressure data could yield important insights into the physiologic events responsible for cardiovascular morbidity. Such information could then be used to develop diagnostic tests that identify those people at highest risk and thus who might especially benefit from intervention. This would be of potentially great public health importance, given the prevalence of SDB and the availability of treatments for SDB.

DESIGN NARRATIVE:

The investigators used the computerized database of the Wisconsin Sleep Cohort to answer the following specific questions. What were the physiologic characteristics of SDB events in the non-clinical population in terms of severity, high airway resistance, obstructive and central components and associated after-effects on EEG arousal and ventilatory overshoots? Did these important elements of the SDB event change as SDB progressed over time? Did the ventilatory or cardiovascular consequences of apnea or hypopnea and its immediate aftermath determine the likelihood of subsequent sleep-disordered breathing events? 2. What were the immediate and long-term cardiovascular consequences of sleep-disordered breathing events; what characteristics of these SDB events (such as oxygen desaturation, arousal, ventilatory overshoot airway resistance, etc.) determined the cardiovascular responses and consequences? 3. What was the effect of aging on SDB and its sequelae as studied in the truly healthy elderly? 4. What role did anatomical characteristics of the upper airway play in determining the frequency and severity and type of sleep-disordered breathing? Did these anatomical determinants differ in the general non-clinical population versus the obstructive sleep apnea (OSA) population? ... in the obese versus the non-obese?

Organization responded that the study is non-FDAAA applicable and they do not accept transfer to their organization.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-04; Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Dempsey — University of Wisconsin, Madison

REFERENCES:
- [Background] Dempsey JA, Skatrud JB, Jacques AJ, Ewanowski SJ, Woodson BT, Hanson PR, Goodman B. Anatomic determinants of sleep-disordered breathing across the spectrum of clinical and nonclinical male subjects. Chest. 2002 Sep;122(3):840-51. doi: 10.1378/chest.122.3.840. PMID 12226022